CLINICAL TRIAL: NCT01056276
Title: Phase II Study for the Evaluation of Bendamustine, Bortezomib and Dexamethasone (BBD) in the First-Line Treatment of Patients With Multiple Myeloma Who Are Not Candidates for High Dose Chemotherapy
Brief Title: Study to Evaluate the Combination of Bendamustine, Bortezomib and Dexamethasone (BBD) in the First-Line Treatment of Patients With Multiple Myeloma Who Are Not Candidates for High Dose Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI MM 23
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bendamustine; Bortezomib; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Bendamustine, Bortezomib,and Dexamethasone for 8 cycles or 2 cycles beyond a confirmed complete response, assessed by IMWG criteria. Patients with stable disease and no intolerable toxicity may continue maintenance therapy with Bortezomib and Dexamethasone until disease progression or intolerable toxicity.
  Interventions: Drug: Bendamustine; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bendamustine — Treatment: 80 mg/m2 via intravenous (IV) Days 1 and 2; repeat cycles every 28-days for 8 cycles or 2 cycles beyond confirmed complete response.
  Other Names: Treanda
Drug: Bortezomib — 1.3 mg/m2 IV Days 1, 8, 15; repeat cycles every 28-days for 8 cycles or 2 cycles beyond confirmed complete response.
  Maintenance: 1.3 mg/m2 IV or SQ Days 1, 15
  Other Names: Velcade
Drug: Dexamethasone — 20 mg orally (PO) Days 1, 2, 8, 9, 15, 16 every 28-days for 8 cycles or 2 cycles beyond confirmed complete response, Maintenance: 20 mg PO Days 1, 15

SUMMARY:
In this study, investigators will evaluate the activity of bendamustine, bortezomib and dexamethasone (BBD). This regimen combines 3 agents with high activity in multiple myeloma, with different mechanisms of action and non-overlapping toxicities.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy, tolerability, and toxicity of bendamustine, bortezomib, and dexamethasone (BBD) as first-line treatment of multiple myeloma (MM) patients who are transplant ineligible or who are not candidates for high dose chemotherapy. Eligible patients will receive protocol treatment for up to 34 weeks plus the screening period (up to 2 weeks). Response assessments will occur every 4 weeks and confirmed using the International Myeloma Working Group Uniform Response Criteria. Patients having an objective response or stable disease will continue to maintenance therapy until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must meet the Durie and Salmon criteria for initial diagnosis of multiple myeloma.
2. Previously histologically confirmed, multiple myeloma with indication for therapy including one of the following:

   * Hemoglobin <10 g/dl or 2 g/dl below normal
   * Serum calcium >11.5 mg/dl
   * Creatinine >2 mg/dl
   * Lytic bone lesions or severe osteopenia
   * Extramedullary plasmacytomas
3. Patients should not be considered candidates for high dose therapy/autologous stem cell transplantation due to coexistent medical conditions, advanced age, poor performance status, refusal of high dose chemotherapy, or other reasons as judged by the patient and/or physician.
4. ECOG Performance Status 0-2.
5. WBC ≥3000/mL; ANC ≥1000/mL; platelets ≥50,000/mL (patients with platelets ≥30,000/mL are eligible if thrombocytopenia is felt to be due to extensive bone marrow involvement with myeloma).
6. Patients with adequate organ function as measured by:

   Renal: Serum creatinine <2.0 mg/dL or a calculated or measured creatinine clearance of >30 mL/minute.

   Hepatic: Total bilirubin < 1.5 x ULN and ALT and AST <2.5 x the ULN (<5 x ULN for patients with liver involvement).
7. Patients must have measurable or evaluable disease. In patients with disease limited to bone and bone marrow, serial paraprotein measurements are acceptable for evaluable disease.
8. Patients must be accessible for treatment and follow-up procedures.
9. Male or female patients 18 years of age or older.
10. Patients must provide written informed consent prior to receiving protocol therapy.
11. Women of childbearing potential must agree to use a medically acceptable method of birth control(e.g., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study and for 12 months after their last dose of rituximab. Men must use an acceptable form/method of contraception for the duration of treatment and for 3 months after the end of treatment.
12. Patients must be able to understand the nature of this study and give written informed consent.

Exclusion Criteria:

1. Previous therapy for multiple myeloma with the exception of an initial 4-day course of pulsed dexamethasone.
2. Patients with ≥NCI CTCAE v4.0 grade 2 peripheral neuropathy ≤14 days prior to study enrollment.
3. Treatment with investigational agent(s) ≤14 days prior to study enrollment.
4. Active infection or infection requiring intravenous antibiotic treatment at the time of accrual.
5. Known to be HIV positive (HIV test is not required for participation in the trial).
6. Patients with class III/IV cardiac problems as defined by the New York Heart Association (NYHA)criteria:

   * History of uncontrolled or symptomatic angina
   * History of arrhythmias requiring medications, or clinically significant, with the exception of asymptomatic atrial fibrillation requiring anticoagulation
   * Myocardial infarction < 6 months from study entry
   * Uncontrolled or symptomatic congestive heart failure
   * Ejection fraction below the institutional normal limit
   * Any other cardiac condition that, in the opinion of the treatment physician, would make this protocol unreasonably hazardous for the patient
   * Uncontrolled hypertension (systolic blood pressure [BP] >180 or diastolic BP >100mm Hg)or uncontrolled cardiac arrhythmias.
   * Prior to study entry, any ECG abnormality at Screening must be documented by the investigator as not medically relevant.
7. Other serious medical conditions or psychiatric illness that would potentially interfere with patient participation in this trial.
8. A second malignancy, other than basal cell carcinoma of the skin or in situ carcinoma of the cervix,unless the tumor was treated with curative intent at least 2 years previously or low-risk prostate cancer after curative therapy.
9. Known hypersensitivity to bortezomib, boron, or mannitol.
10. Female patient is pregnant or lactating. Confirmation that female patients of childbearing potential are not pregnant must be established by a negative serum pregnancy test ≤7 days prior to start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-05; Primary Completion 2015-08 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Berdeja, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (13):
- United States (13):
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Hematology Oncology Clinic, LLP, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Oncology Hematology Care Inc., Cincinnati, Ohio
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Leading Edge Research, PA, Arlington, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Peninsula Cancer Institute, Newport News, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2010 and May 2014, 59 patients with transplant-ineligible Multiple Myeloma (MM) were enrolled at 9 investigational sites in the U.S. The original treatment plan was modified during the trial to decrease intensity but increase treatment duration. Of 59 enrolled patients, 18 were treated on the initial regimen; 41 on the modified plan.
Groups:
- Original BBD Regimen: Bendamustine, Bortezomib,and Dexamethasone (BBD) every 28 days for 8 cycles or 2 cycles beyond a confirmed complete response, assessed by International Myeloma Working Group (IMWG) Uniform Response Criteria. No maintenance therapy.
  Bendamustine: 80 mg/m2 via intravenous (IV) Days 1 and 4 Bortezomib: 1.3 mg/m2 IV Days 1, 4, 8, 11 Dexamethasone: 40 mg orally (PO) Days 1, 2, 3, 4
- Modified BBD Regimen: Bendamustine, Bortezomib,and Dexamethasone (BBD) every 28 days for 8 cycles or 2 cycles beyond a confirmed complete response, assessed by International Myeloma Working Group (IMWG) Uniform Response Criteria criteria. Patients with stable disease and no intolerable toxicity may continue maintenance therapy with Bortezomib and Dexamethasone every 28 days for 4 cycles. After cycle 4, dexamethasone may be discontinued at the physician's discretion.
  Treatment:
  Bendamustine: 80 mg/m2 via intravenous (IV) Days 1 and 2 Bortezomib: 1.3 mg/m2 IV Days 1, 8, 15 Dexamethasone: 20 mg orally (PO) Days 1, 2, 8, 9, 15,16
  Maintenance:
  Bortezomib: 1.3 mg/m2 IV or SQ Days 1, 15 Dexamethasone: 20 mg PO Days 1, 15
Period: Treatment Period-Cycles 1-8
Arm/Group | Original BBD Regimen | Modified BBD Regimen
Started | 18 | 41
Completed | 5 | 33
Not Completed | 13 | 8
Not completed — Toxicity | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Disease Progression | 2 | 2
Not completed — Intercurrent Illness | 1 | 2
Not completed — Physician Decision | 3 | 0
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Maintenance Therapy
Arm/Group | Original BBD Regimen | Modified BBD Regimen
Started | 0 (Original regimen did not include maintenance therapy.) | 28 (5 patients completed 8 cycles but did not have maintenance therapy.)
Completed | 0 | 0 (14 patients are continuing maintenance therapy.)
Not Completed | 0 | 28
Not completed — Toxicity | 0 | 2
Not completed — Progressive Disease | 0 | 9
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Intercurrent Illness | 0 | 1
Not completed — Continuing maintenance therapy | 0 | 14

BASELINE CHARACTERISTICS:
Population: All patients enrolled in either the original treatment regimen or the modified treatment regimen.
Groups:
- Total: Total of all reporting groups
Arm/Group | Original BBD Regimen | Modified BBD Regimen | Total
Number analyzed (Participants) | 18 | 41 | 59
Age, Continuous [Median (Full Range); unit: years] | 75 [55 to 81] | 75 [45 to 89] | 75 [45 to 89]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  female | 5 | 14 | 19
  male | 13 | 26 | 39
  unknown | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Black/African American | 3 | 10 | 13
  Caucasian | 14 | 27 | 41
  White | 0 | 2 | 2
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 41 | 59

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Defined as the percent of patients having a complete response (CR) to treatment, assessed using the International Myeloma Working Group (IMWG) Uniform Response Criteria. CR=disappearance of soft tissue plasmacytomas and 5% or less plasma cells in bone marrow.
Time Frame: every 8 weeks for approximately 48 months
Population: All patients evaluable for response.
Measure: Number; unit: percentage of participants
Groups:
- Original BBD Regimen: Bendamustine, Bortezomib,and Dexamethasone (BBD) every 28 days for 8 cycles or 2 cycles beyond a confirmed complete response, assessed by International Myeloma Working Group (IMWG) Uniform Response Criteria criteria. No maintenance therapy.
  Bendamustine: 80 mg/m2 via intravenous (IV) Days 1 and 4 Bortezomib: 1.3 mg/m2 IV Days 1, 4, 8, 11 Dexamethasone: 40 mg orally (PO) Days 1, 2, 3, 4
- Modified BBD Regimen: Bendamustine, Bortezomib,and Dexamethasone (BBD) every 28 days for 8 cycles or 2 cycles beyond a confirmed complete response, assessed by International Myeloma Working Group (IMWG) Uniform Response Criteria criteria. Patients with stable disease and no intolerable toxicity may continue maintenance therapy with Bortezomib and Dexamethasone every 28 days for 4 cycles. After cycle 4, dexamethasone may be discontinued at the physician's discretion.
  Bendamustine: 80 mg/m2 via intravenous (IV) Days 1 and 2 Bortezomib: 1.3 mg/m2 IV Days 1, 8, 15 Dexamethasone: 20 mg orally (PO) Days 1, 2, 8, 9, 15,16
  Maintenance:
  Bortezomib: 1.3 mg/m2 IV or SQ Days 1, 15 Dexamethasone: 20 mg PO Days 1, 15
Arm/Group | Original BBD Regimen | Modified BBD Regimen
Number analyzed (Participants) | 17 | 39
percentage of participants | 0 | 13

2. Primary Outcome: Number of Patients Who Experienced Serious and Non-serious Adverse Events
Description: All serious adverse events (SAEs) and non-serious adverse events (AEs) were assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0, and were collected from start of study treatment until 30 days after last dose of study medication. Refer to the Adverse Event module for specific terms.
Time Frame: approximately 36 weeks
Population: All patients who received at least one dose of BBD treatment.
Measure: Number; unit: participants
Arm/Group | Original BBD Regimen | Modified BBD Regimen
Number analyzed (Participants) | 18 | 41
participants
  SAEs | 7 | 17
  AEs | 18 | 38

3. Secondary Outcome: Progression Free Survival
Description: Defined as the interval of time (in months) that patient are alive from date of first protocol treatment to date of documented tumor progression or date of death from any cause. Progressive disease, assessed according to International Myeloma Working Group Uniform Response Criteria, is defined as at least a 25% increase from the nadir in any one of the following criteria: serum M-protein, urine M-protein, or bone marrow plasma cell percentage of 10% or greater.
Time Frame: every 8 weeks for up to 48 months
Measure: Median (Full Range); unit: months
Groups:
- Modified BBD Regimen: Bendamustine, Bortezomib,and Dexamethasone (BBD) every 28 days for 8 cycles or 2 cycles beyond a confirmed complete response, assessed by International Myeloma Working Group (IMWG) Uniform Response Criteria. Patients with stable disease and no intolerable toxicity may continue maintenance therapy with Bortezomib and Dexamethasone every 28 days for 4 cycles. After cycle 4, dexamethasone may be discontinued at the physician's discretion.
  Treatment:
  Bendamustine: 80 mg/m2 via intravenous (IV) Days 1 and 2 Bortezomib: 1.3 mg/m2 IV Days 1, 8, 15 Dexamethasone: 20 mg orally (PO) Days 1, 2, 8, 9, 15,16
  Maintenance:
  Bortezomib: 1.3 mg/m2 IV or SQ Days 1, 15 Dexamethasone: 20 mg PO Days 1, 15
Arm/Group | Original BBD Regimen | Modified BBD Regimen
Number analyzed (Participants) | 17 | 39
months | 11.1 [5.5 to 16.3] | 18.9 [14.1 to 31.8]

4. Secondary Outcome: Overall Survival
Description: Defined as the interval of time, in months, from first study treatment until the earlier of the date of death or date last known alive.
Time Frame: every 4 weeks until progressive disease then every 12 weeks, projected 48 months
Population: All patients evaluable for response.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- BBD Treatment: Bendamustine, Bortezomib,and Dexamethasone (BBD) every 28 days for 8 cycles or 2 cycles beyond a confirmed complete response, assessed by International Myeloma Working Group (IMWG) Uniform Response Criteria. Patients with stable disease and no intolerable toxicity may continue maintenance therapy with Bortezomib and Dexamethasone every 28 days for 4 cycles. After cycle 4, dexamethasone may be discontinued at the physician's discretion.
  Treatment:
  Bendamustine: 80 mg/m2 via intravenous (IV) Days 1 and 2 Bortezomib: 1.3 mg/m2 IV Days 1, 8, 15 Dexamethasone: 20 mg orally (PO) Days 1, 2, 8, 9, 15,16
  Maintenance:
  Bortezomib: 1.3 mg/m2 IV or SQ Days 1, 15 Dexamethasone: 20 mg PO Days 1, 15
Arm/Group | Original BBD Regimen | BBD Treatment
Number analyzed (Participants) | 17 | 39
months | NA [NA to NA] — Median overall survival has not been reached. | NA [NA to NA] — Median overall survival has not been reached..

5. Secondary Outcome: Overall Response Rate
Description: The number of patients with observed complete or partial response (CR or PR) assessed by International Myeloma Working Group (IMWG) Uniform Response Criteria. PR=50% or greater reduction from baseline in serum M-protein and 90% or greater reduction from baseline in 24-hour urinary M-protein.
Time Frame: every 4 weeks for approximately 2 years
Population: All patients evaluable for response.
Measure: Number; unit: participants
Groups:
- Originl BBD Regimen: Bendamustine, Bortezomib,and Dexamethasone (BBD) every 28 days for 8 cycles or 2 cycles beyond a confirmed complete response, assessed by International Myeloma Working Group (IMWG) Uniform Response Criteria. No maintenance therapy.
  Bendamustine: 80 mg/m2 via intravenous (IV) Days 1 and 4 Bortezomib: 1.3 mg/m2 IV Days 1, 4, 8, 11 Dexamethasone: 40 mg orally (PO) Days 1, 2, 3, 4
Arm/Group | Originl BBD Regimen | Modified BBD Regimen
Number analyzed (Participants) | 17 | 39
participants
  CR | 0 | 5
  PR | 5 | 8

ADVERSE EVENTS:
Time Frame: every 4 weeks for up to 32 weeks on the Original BBD Regimen, or up to 2 years on the Modified BBD Regimen
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were collected from day of first dose to 30 days after last dose of study medication and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Arm/Group | Original BBD Regimen | Modified BBD Regimen
Serious Adverse Events (participants affected / at risk) | 7/18 | 17/41
Other Adverse Events (participants affected / at risk) | 18/18 | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Original BBD Regimen (N=18) | Modified BBD Regimen (N=41)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 5 (9)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Salivary duct obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Original BBD Regimen (N=18) | Modified BBD Regimen (N=41)
FATIGUE (General disorders) | 13 | 31
PERIPHERAL NEUROPATHY (Nervous system disorders) | 13 | 28
ANEMIA (Blood and lymphatic system disorders) | 7 | 23
EDEMA (General disorders) | 6 | 21
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 18
CONSTIPATION (Gastrointestinal disorders) | 9 | 18
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 9 | 18
INSOMNIA (Nervous system disorders) | 6 | 17
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 15
DIARRHEA (Gastrointestinal disorders) | 5 | 15
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 15
NEUTROPENIA (Blood and lymphatic system disorders) | 7 | 14
NAUSEA (Gastrointestinal disorders) | 10 | 13
ANOREXIA (Metabolism and nutrition disorders) | 6 | 13
LEUKOPENIA (Blood and lymphatic system disorders) | 8 | 13
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 11
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 10
RASH (Skin and subcutaneous tissue disorders) | 1 | 10
MYALGIA (Musculoskeletal and connective tissue disorders) | 12 | 10
ASTHENIA (General disorders) | 2 | 10
FEVER (General disorders) | 2 | 9
DIZZINESS (Nervous system disorders) | 4 | 9
NEUROPATHY (Nervous system disorders) | 0 | 8
PAIN (General disorders) | 1 | 7
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 2 | 7
HYPERTENSION (Vascular disorders) | 1 | 6
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 6
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 6
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 3 | 6
DYSPEPSIA (Gastrointestinal disorders) | 4 | 6
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 4 | 6
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 5
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 5
WEIGHT LOSS (Investigations) | 1 | 5
DYSGEUSIA (Nervous system disorders) | 2 | 5
DEPRESSION (Psychiatric disorders) | 3 | 5
HYPOTENSION (Vascular disorders) | 3 | 5
TASTE ALTERATION (Nervous system disorders) | 3 | 5
CATARACT (Eye disorders) | 0 | 4
CHEST CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 4
INFECTION (Infections and infestations) | 0 | 4
CREATININE LEVELS INCREASED (Investigations) | 1 | 4
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 | 4
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 4
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 4
ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 3
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 3
BRONCHIAL INFECTION (Infections and infestations) | 0 | 3
BRUISING (Injury, poisoning and procedural complications) | 0 | 3
DYSPHAGIA (Gastrointestinal disorders) | 0 | 3
HEARING IMPAIRED (Ear and labyrinth disorders) | 0 | 3
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3
SKIN CHANGES (Skin and subcutaneous tissue disorders) | 0 | 3
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 | 3
URINARY TRACT INFECTION (Renal and urinary disorders) | 0 | 3
CHEST PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 3
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 3
NASAL DRAINAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 3
PARESTHESIA (Nervous system disorders) | 1 | 3
GAIT DISTURBANCE (General disorders) | 2 | 3
DEHYDRATION (Metabolism and nutrition disorders) | 5 | 3
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 2
BLURRED VISION (Eye disorders) | 1 | 2
FALL (Injury, poisoning and procedural complications) | 1 | 2
FLU LIKE SYMPTOMS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 | 2
THRUSH (Infections and infestations) | 1 | 2
CHILLS (General disorders) | 2 | 2
VOMITING (Gastrointestinal disorders) | 2 | 2
HEADACHE (Nervous system disorders) | 3 | 2
HERPES ZOSTER (Infections and infestations) | 8 | 2
URINARY FREQUENCY (Renal and urinary disorders) | 2 | 1
ALLERGIC REACTION (Immune system disorders) | 3 | 1
MUCOSITIS (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.